CLINICAL TRIAL: NCT05900609
Title: Gut Health Enhancement by Eating Favourable Food
Acronym: GEEFomjebuik
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VU University of Amsterdam (Other)
Collaborators: Wageningen University and Research (Other); Maag Lever Darm Stichting (Other); Cidrani (Unknown); WholeFiber (Unknown); Keep Food Simple (Unknown)
Responsible Party: Principal Investigator, Remco Kort, Professor doctor, VU University of Amsterdam
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: NL83652.028.23
Record Dates: First submitted 2023-04-03; First posted 2023-06-12 (Actual); Last update posted 2025-07-08 (Actual); Status verified 2025-07

CONDITIONS: Microbial Colonization
Keywords: Fiber; Fermented food; Immune system; Microbiota
MeSH Terms: conditions — Communicable Diseases | interventions — Kombucha Tea

STUDY DESIGN:
Intervention Model Description: The study applies a randomized, parallel design of 8 weeks (+ follow-up after 3 months)
Masking Description: This study is partially blinded, study participants in the fiber and fermented group will be informed about their intervention after randomization. However, the control group will remain blind throughout the intervention period. Furthermore, participants are not made aware of the different types of intervention before start or during the intervention period. This is done to prevent any adjustments of their diets based on the advices in the other groups and to ensure that the control group stays blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Fiber arm (Experimental): Subjects receive dietary guidelines, to increase their fiber intake. Additionally, during the last 6 weeks of the intervention period subjects receive a study product containing 8,5 grams fiber per day.
  Additionally, subjects receive general guidelines about the effect of nutrition on the gut microbiome.
  Interventions: Dietary Supplement: WholeFiber
- Fermented food arm (Experimental): Subjects receive dietary guidelines, to increase their intake of fermented foods.
  Additionally, during the last 6 weeks of the intervention period subjects receive a study product of 17 millilitres concentrated kombucha per day.
  Additionally, subjects receive general guidelines about the effect of nutrition on the gut microbiome.
  Interventions: Dietary Supplement: Kombucha
- Control (Placebo Comparator): Subjects receive general guidelines about the effect of nutrition on the gut microbiome.
  Additionally, during the last 6 weeks of the intervention period subjects receive a placebo product of 10 grams maltodextrin per day.
  Interventions: Dietary Supplement: Maltodextrin DE19/21

INTERVENTIONS:
Dietary Supplement: WholeFiber — WholeFiberTM is a product with high levels of prebiotic dietary fibers (~85%) mainly consisting of inulin, and some pectin, hemi-cellulose and cellulose that is derived from the root vegetable, chicory roots.
  Fiber guidelines:
  Subjects receive a booklet with recipes high in fiber. Subjects are recommended to use 2 recipes + 2 snacks per day. Estimated average intake via the recipes in the recipe booklet is 24 grams/day.
  General guidelines on nutrition and microbiome:
  Subjects receive a link to a website with general recommendations to positively alter the gut microbiome (website Voedingscentrum and Dutch Digestive Foundation).
  Other Names: Chicory roots
  Arms: Fiber arm
Dietary Supplement: Kombucha — The kombucha is produced by a minimum three-month long fermentation process. It is a live fermented herbal drink essence, without refined sugar, and an unpasteurized, organic product.
  Fermented food guidelines:
  Study participants in the fermented foods arm are asked to use 3 additional servings of fermented food per day, using the fermented food list / recipe booklet.
  General guidelines on nutrition and microbiome:
  Subjects receive a link to a website with general recommendations to positively alter the gut microbiome (website Voedingscentrum and Dutch Digestive Foundation).
  Other Names: Fermented tea
  Arms: Fermented food arm
Dietary Supplement: Maltodextrin DE19/21 — Maltodextrin DE19/21 is a digestible carbohydrate, that is completely digested and does not reach the colon, which makes it a suitable placebo dietary compound and the reason why it is frequently used in comparable studies.
  General guidelines on nutrition and microbiome:
  Subjects receive a link to a website with general recommendations to positively alter the gut microbiome (website Voedingscentrum and Dutch Digestive Foundation).
  Arms: Control

SUMMARY:
Within the GEEF om je buik study the effects of an 8-week intervention with either a diet rich in fiber or fermented food on the gut microbiota will be investigated.

DETAILED DESCRIPTION:
This study is a randomized controlled trial (RCT) with three intervention groups (high dietary fiber group (HDF), high fermented foods group (HFF), and a control group (CG)). The total duration of the study is 5 months and consists of an 8-week intervention (2-week ramp up period with dietary guidelines, followed by 6-week period with dietary guidelines + additional consumption of study products) and a follow-up after 3 months. In total 147 subjects will be included.

ELIGIBILITY:
Inclusion Criteria:

* Men and Women, aged ≥18 - ≤70 years;
* Being able to read and speak Dutch;
* Willing to keep a stable dietary pattern throughout the study, apart from the dietary advice in the study;
* Having a smartphone compatible with the Lifedata or PocketQ app to fill out the daily questionnaires.

Exclusion Criteria:

* Having a disease or medical condition which can influence the study results such as diabetes, cancer, diagnosed irritable bowel syndrome, renal disease, liver enzyme abnormality, malignant neoplasm, or a history of inflammatory diseases (such as multiple sclerosis, rheumatoid arthritis, and inflammatory bowel disease);
* Having a history of intestinal surgery that might interfere with study outcomes (this does not include an appendectomy or cholecystectomy);
* Average dietary fiber intake of ≥18 gram (women) or ≥22 gram (men) per day, according to the fiber screen questionnaire (see F1 questionnaires);
* More than 3 servings of fermented foods per day as assessed with the fermented food frequency questionnaire (see F1 questionnaires);
* Having a Body Mass Index (BMI) of ≥ 30 kg/m2 (self-reported);
* Currently following a strict diet and unwilling or unable to change; for example, a gluten free diet or a "crash diet" using meal substitutes;
* Specific food allergies that interfere with dietary intervention (for example, gluten, lactose, etc);
* Use of prebiotics, probiotics and/or synbiotics (this should be stopped 4 weeks before the start of the study) and use of fiber supplements;
* Use of antibiotic treatment less than 3 months before start of the study and/or use of antibiotics during the study;
* Use of medication that can interfere with the study outcomes, as judged by the medical supervisor;
* Alcoholic use of ≥14 (women) or ≥28 (men) glasses of alcoholic beverages per week;
* Use of soft or hard drugs (should be stopped at least 4 weeks before start of the study);
* Being pregnant or lactating;
* Participation in another clinical trial at the same time;
* Student or employee working at either Food, Health and Consumer Research from Wageningen Food and Biobased Research, Microbiology at VU, the MLDS, at WholeFiber, Keep Food Simple or at Cidrani;
* Unable to follow or comply to study rules.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 146 (Actual)
Dates: Start 2023-05-22 (Actual); Primary Completion 2023-11-26 (Actual); Study Completion 2024-03-06 (Actual)

PRIMARY OUTCOMES:
Microbiota diversity | Baseline (week 0)
  Microbial richness (ASV) using 16s rRNA
Microbiota diversity | End ramp-up (week 2)
  Microbial richness (ASV) using 16s rRNA
Microbiota diversity | End intervention (week 8)
  Microbial richness (ASV) using 16s rRNA

SECONDARY OUTCOMES:
Gut microbiota composition | Baseline (week 0)
  16s rRNA
Gut microbiota composition | End ramp-up (week 2)
  16s rRNA
Gut microbiota composition | End intervention (week 8)
  16s rRNA
Carbohydrate Active Enzymes (CAZymes) | Baseline (week 0)
  Relative abundance of CAZymes using shotgun metagenomic sequencing
Carbohydrate Active Enzymes (CAZymes) | End ramp-up (week 2)
  Relative abundance of CAZymes using shotgun metagenomic sequencing
Carbohydrate Active Enzymes (CAZymes) | End intervention (week 8)
  Relative abundance of CAZymes using shotgun metagenomic sequencing
92 inflammatory serum proteins | Baseline (week 0)
  92 protein biomarkers proteins associated with inflammatory and immune response processes measured in dried blood spots using the Olink target 96 panels. Expressed as normalized protein expression (NPX).
92 inflammatory serum proteins | End ramp-up (week 2)
  92 protein biomarkers proteins associated with inflammatory and immune response processes measured in dried blood spots using the Olink target 96 panels. Expressed as normalized protein expression (NPX).
92 inflammatory serum proteins | End intervention (week 8)
  92 protein biomarkers proteins associated with inflammatory and immune response processes measured in dried blood spots using the Olink target 96 panels. Expressed as normalized protein expression (NPX).
Dietary intake | Baseline (week 0)
  Average intake of fiber, fermented foods and macronutrients using the Traqq app
Dietary intake | End ramp-up (week 2)
  Average intake of fiber, fermented foods and macronutrients using the Traqq app
Dietary intake | End intervention (week 8)
  Average intake of fiber, fermented foods and macronutrients using the Traqq app
Dietary intake | End follow-up (5 months)
  Average intake of fiber, fermented foods and macronutrients using the Traqq app
Gastrointestinal complaints | Daily during intervention (week 0 - week 8)
  Likert-point scale (scores 0 - 10), for bloating, flatulence and abdominal pain. A higher score means more bloating, flatulence and abdominal pain.
Stool frequency | Daily during intervention (week 0 - week 8)
  Frequency of bowel movement per day
Stool consistency | Daily during intervention (week 0 - week 8)
  Consistency per stool, based on Bristol Stool Score (type 1 -7). Scores 1-7. A higher score means more loose / watery stool.
Abundance of Prevotella | Baseline (week 0)
  Based on a faecal smear image, using MicrobeLink tool from HORAIZON (AI, machine learning).
Abundance of Prevotella | End ramp-up (week 2)
  Based on a faecal smear image, using MicrobeLink tool from HORAIZON (AI, machine learning).
Abundance of Prevotella | End intervention (week 8)
  Based on a faecal smear image, using MicrobeLink tool from HORAIZON (AI, machine learning).
Abundance of Bacteroides | Baseline (week 0)
  Based on a faecal smear image, using MicrobeLink tool from HORAIZON (AI, machine learning).
Abundance of Bacteroides | End ramp-up (week 2)
  Based on a faecal smear image, using MicrobeLink tool from HORAIZON (AI, machine learning).
Abundance of Bacteroides | End intervention (week 8)
  Based on a faecal smear image, using MicrobeLink tool from HORAIZON (AI, machine learning).
Ratio of Prevotella/Bacteroides | Baseline (week 0)
  Based on a faecal smear image, using MicrobeLink tool from HORAIZON (AI, machine learning).
Ratio of Prevotella/Bacteroides | End ramp-up (week 2)
  Based on a faecal smear image, using MicrobeLink tool from HORAIZON (AI, machine learning).
Ratio of Prevotella/Bacteroides | End intervention (week 8)
  Based on a faecal smear image, using MicrobeLink tool from HORAIZON (AI, machine learning).
Microbial alpha diversity | Baseline (week 0)
  Based on a faecal smear image, using MicrobeLink tool from HORAIZON (AI, machine learning).
Microbial alpha diversity | End ramp-up (week 2)
  Based on a faecal smear image, using MicrobeLink tool from HORAIZON (AI, machine learning).
Microbial alpha diversity | End intervention (week 8)
  Based on a faecal smear image, using MicrobeLink tool from HORAIZON (AI, machine learning).
Transit time | Baseline (week 0)
  Using blue dye method (two blue muffins)
Transit time | End ramp-up (week 2)
  Using blue dye method (two blue muffins)
Transit time | End intervention (week 8)
  Using blue dye method (two blue muffins)
Sleep quality | Baseline (week 0)
  Athens insomnia scale. Score range: 0-28 points. Higher score means worse outcome.
Sleep quality | End ramp-up (week 2)
  Athens insomnia scale. Score range: 0-28 points. Higher score indicates worse sleep quality.
Sleep quality | End intervention (week 8)
  Athens insomnia scale. Score range: 0-28 points. Higher score indicates worse sleep quality.
Sleep quality | End follow-up (5 months)
  Athens insomnia scale. Score range: 0-28 points. Higher score indicates worse sleep quality.
Digestion associated Quality of Life | Baseline (week 0)
  Digestion associated Quality of Life (DQLQ) questionnaire. Score range: 0-9. Higher score indicates worse digestion associated quality of life.
Digestion associated Quality of Life | End ramp-up (week 2)
  Digestion associated Quality of Life (DQLQ) questionnaire. Score range: 0-9. Higher score indicates worse digestion associated quality of life.
Digestion associated Quality of Life | End intervention (week 8)
  Digestion associated Quality of Life (DQLQ) questionnaire. Score range: 0-9. Higher score indicates worse digestion associated quality of life.
Digestion associated Quality of Life | End follow-up (5 months)
  Digestion associated Quality of Life (DQLQ) questionnaire. Score range: 0-9. Higher score indicates worse digestion associated quality of life.
Well-being | Baseline (week 0)
  World Health Organisation (WHO)-Five Well-Being Index (WHO-5) questionnaire. Raw score ranges from 0-25. Final score is calculated by multiplying the raw score by 4. Final score range 0-100. Higher score indicates better well-being.
Well-being | End ramp-up (week 2)
  World Health Organisation (WHO)-Five Well-Being Index (WHO-5) questionnaire. Raw score ranges from 0-25. Final score is calculated by multiplying the raw score by 4. Final score range 0-100. Higher score indicates better well-being.
Well-being | End intervention (week 8)
  World Health Organisation (WHO)-Five Well-Being Index (WHO-5) questionnaire. Raw score ranges from 0-25. Final score is calculated by multiplying the raw score by 4. Final score range 0-100. Higher score indicates better well-being.
Well-being | End follow-up (5 months)
  World Health Organisation (WHO)-Five Well-Being Index (WHO-5) questionnaire. Raw score ranges from 0-25. Final score is calculated by multiplying the raw score by 4. Final score range 0-100. Higher score indicates better well-being.
Subjective health (perception and awareness) | Baseline (week 0)
  A 2-item questionnaire, which assesses how healthy participants perceive their own health and diet. Score range: 2 - 14, higher scores mean a higher subjective health
Subjective health (perception and awareness) | End intervention (week 8)
  A 2-item questionnaire, which assesses how healthy participants perceive their own health and diet. Score range: 2 - 14, higher scores mean a higher subjective health
Subjective health (perception and awareness) | End follow-up (5 months)
  A 2-item questionnaire, which assesses how healthy participants perceive their own health and diet. Score range: 2 - 14, higher scores mean a higher subjective health
Intention to stay healthy (perception + awareness) | Baseline (week 0)
  A 3-item questionnaire, which assesses the extent to which participants have the intention to eat healthy. Score range: 3 - 21, higher scores mean more intention to stay healthy
Intention to stay healthy (perception + awareness) | End intervention (week 8)
  A 3-item questionnaire, which assesses the extent to which participants have the intention to eat healthy. Score range: 3 - 21, higher scores mean more intention to stay healthy
Intention to stay healthy (perception + awareness) | End follow-up (5 months)
  A 3-item questionnaire, which assesses the extent to which participants have the intention to eat healthy. Score range: 3 - 21, higher scores mean more intention to stay healthy
Dietary intrinsic motivation (perception + awareness) | Baseline (week 0)
  A validated 6-item questionnaire, which assesses whether someone's motivation to eat healthy comes from within a person. Score range: 6 - 42, higher scores mean a higher intrinsic motivation.
Dietary intrinsic motivation (perception + awareness) | End intervention (week 8)
  A validated 6-item questionnaire, which assesses whether someone's motivation to eat healthy comes from within a person. Score range: 6 - 42, higher scores mean a higher intrinsic motivation.
Dietary intrinsic motivation (perception + awareness) | End follow-up (5 months)
  A validated 6-item questionnaire, which assesses whether someone's motivation to eat healthy comes from within a person. Score range: 6 - 42, higher scores mean a higher intrinsic motivation.
Dietary self-efficacy (perception + awareness) | Baseline (week 0)
  A validated 8-item questionnaire, which assesses the extent to which one feels capable of eating healthy. Score range: 8 - 49, higher scores mean a higher self-efficacy
Dietary self-efficacy (perception + awareness) | End intervention (week 8)
  A validated 8-item questionnaire, which assesses the extent to which one feels capable of eating healthy. Score range: 8 - 49, higher scores mean a higher self-efficacy
Dietary self-efficacy (perception + awareness) | End follow-up (5 months)
  A validated 8-item questionnaire, which assesses the extent to which one feels capable of eating healthy. Score range: 8 - 49, higher scores mean a higher self-efficacy
Self-regulation (perception + awareness) | Baseline (week 0)
  A 5-item questionnaire, which assesses the ability to plan and monitor actions. Score range: 5 - 35, higher scores mean a higher self-regulation
Self-regulation (perception + awareness) | End intervention (week 8)
  A 5-item questionnaire, which assesses the ability to plan and monitor actions. Score range: 5 - 35, higher scores mean a higher self-regulation
Self-regulation (perception + awareness) | End follow-up (5 months)
  A 5-item questionnaire, which assesses the ability to plan and monitor actions. Score range: 5 - 35, higher scores mean a higher self-regulation
Subjective knowledge (perception + awareness) | Baseline (week 0)
  A validated 5-item questionnaire, which assesses how knowledgeable someone feels about nutrition and gut microbiota. Score range: 5 - 35, higher scores mean a higher subjective knowledge
Subjective knowledge (perception + awareness) | End intervention (week 8)
  A validated 5-item questionnaire, which assesses how knowledgeable someone feels about nutrition and gut microbiota. Score range: 5 - 35, higher scores mean a higher subjective knowledge
Subjective knowledge (perception + awareness) | End follow-up (5 months)
  A validated 5-item questionnaire, which assesses how knowledgeable someone feels about nutrition and gut microbiota. Score range: 5 - 35, higher scores mean a higher subjective knowledge

OTHER OUTCOMES:
Body Mass Index (BMI) | Baseline (week 0)
  Weight and height will be combined to report BMI in kg/m^2
Body Mass Index (BMI) | End ramp-up (week 2)
  Weight and height will be combined to report BMI in kg/m^2
Body Mass Index (BMI) | End intervention (week 8)
  Weight and height will be combined to report BMI in kg/m^2
Body Mass Index (BMI) | End follow-up (5 months)
  Weight and height will be combined to report BMI in kg/m^2

CONTACTS AND LOCATIONS:
Overall Officials: Nicole de Wit, PhD, Principal Investigator — Wageningen Food and Biobased Research; Remco Kort, PhD, Principal Investigator — VU University of Amsterdam
Locations (1):
- Stichting Wageningen Research, Wageningen, Gelderland, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wastyk HC, Fragiadakis GK, Perelman D, Dahan D, Merrill BD, Yu FB, Topf M, Gonzalez CG, Van Treuren W, Han S, Robinson JL, Elias JE, Sonnenburg ED, Gardner CD, Sonnenburg JL. Gut-microbiota-targeted diets modulate human immune status. Cell. 2021 Aug 5;184(16):4137-4153.e14. doi: 10.1016/j.cell.2021.06.019. Epub 2021 Jul 12. PMID 34256014
- [Background] David LA, Maurice CF, Carmody RN, Gootenberg DB, Button JE, Wolfe BE, Ling AV, Devlin AS, Varma Y, Fischbach MA, Biddinger SB, Dutton RJ, Turnbaugh PJ. Diet rapidly and reproducibly alters the human gut microbiome. Nature. 2014 Jan 23;505(7484):559-63. doi: 10.1038/nature12820. Epub 2013 Dec 11. PMID 24336217
- [Background] Myhrstad MCW, Tunsjo H, Charnock C, Telle-Hansen VH. Dietary Fiber, Gut Microbiota, and Metabolic Regulation-Current Status in Human Randomized Trials. Nutrients. 2020 Mar 23;12(3):859. doi: 10.3390/nu12030859. PMID 32210176
- [Background] Stiemsma LT, Nakamura RE, Nguyen JG, Michels KB. Does Consumption of Fermented Foods Modify the Human Gut Microbiota? J Nutr. 2020 Jul 1;150(7):1680-1692. doi: 10.1093/jn/nxaa077. PMID 32232406